CLINICAL TRIAL: NCT05897411
Title: Factors That Determine the Responses to Meal Ingestion: Deconditioning of Acquired Food Aversion
Brief Title: Deconditioning of Acquired Food Aversion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR(AG)338/2016N
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: meal ingestion; postprandial responses; hedonic sensations; homeostatic sensations; deconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deconditioning (Experimental)
  Interventions: Behavioral: Unmasking previous conditioning procedure
- Sham deconditioning (Sham Comparator)
  Interventions: Behavioral: No unmasking of previous conditioning

INTERVENTIONS:
Behavioral: Unmasking previous conditioning procedure — An explanation of the method for aversive conditioning of the comfort meal (masked administration of the meal with a high fat supplement) will be provided.
  Arms: Deconditioning
Behavioral: No unmasking of previous conditioning — An explanation of the method for aversive conditioning of the comfort meal (masked administration of the meal with a high fat supplement) will not be provided.
  Arms: Sham deconditioning

SUMMARY:
Background. Aversive conditioning impairs the rewarding value of a comfort meal.

Our aim is to demonstrate the potential effect of deconditioning to reverse aversive conditioning and restore the hedonic postprandial response.

Methods: A sham-controlled, randomised, parallel, single-blind study will be performed on 12 healthy women (6 per group). The rewarding value of a comfort meal will be measured at initial exposure, after aversive conditioning (masked administration of the same meal with a high-fat content) and after a deconditioning intervention (unmasking the aversive conditioning paradigm in the deconditioning group vs sham intervention in the control group). Digestive well-being (primary outcome) will be measured every 10 min before and 60 min after ingestion using graded scales. The effect of deconditioning (change from aversive conditioning to deconditioning) will be compared to sham deconditioning in the control group.

Expected results: The comfort meal at first exposure will induce a pleasant postprandial experience, which will be impaired by aversive conditioning; this effect will be reverted by deconditioning and the hedonic value of the comfort meal will be restored.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Difference in postprandial digestive well-being before and after deconditioning | 120 minutes
  Change in digestive well-being measured by a 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation) in response to a probe meal before and after deconditioning.
Difference in postprandial fullness sensation before and after conditioning | 120 minutes
  Change in fullness sensation by a 10 cm scale graded from 0 (not at all) to 10 (very much) in response to a probe meal before and after conditioning.
Change in postprandial mood before and after conditioning | 120 minutes
  Change in mood measured by a 10 cm scale graded from -5 (negative) to +5 (positive) in response to a probe meal before and after conditioning.
Change in postprandial hunger/satiety before and after conditioning | 120 minutes
  Change in mood measured by a 10 cm scale graded from -5 (extremely hungry) to +5 (completely satiate) in response to a probe meal before and after conditioning.
Change in postprandial discomfort before and after conditioning | 120 minutes
  Change in the sensation of discomfort by a 10 cm scale graded from 0 (not at all) to 10 (very much) in response to a probe meal before and after conditioning

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nieto A, Livovsky DM, Azpiroz F. Conditioning by a Previous Experience Impairs the Rewarding Value of a Comfort Meal. Nutrients. 2023 May 9;15(10):2247. doi: 10.3390/nu15102247. PMID 37242129
- [Derived] Nieto A, Livovsky DM, Azpiroz F. Reversal of Conditioned Food Aversion Using a Cognitive Intervention: A Sham-Controlled, Randomized, Parallel Study. Nutrients. 2023 Nov 29;15(23):4962. doi: 10.3390/nu15234962. PMID 38068820